CLINICAL TRIAL: NCT04898946
Title: Serological Response to mRNA and Inactivated COVID-19 Vaccine in Health Care Workers in Hong Kong
Status: Completed | Type: Observational
Sponsor: Hong Kong Sanatorium & Hospital (Industry)
Responsible Party: Principal Investigator, Dr. Jonpaul ST Zee, Specialist in Infectious Disease, Hong Kong Sanatorium & Hospital
Other Study IDs: Covid-19 Vaccine Antibody
Record Dates: First submitted 2021-05-20; First posted 2021-05-24 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Covid-19 Vaccine
MeSH Terms: interventions — sinovac COVID-19 vaccine; BNT162 Vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- BNT162b2: Subjects who receive mRNA vaccine BNT162b2.
  Interventions: Biological: BNT162b2 Vaccine
- CoronaVac: Subjects who receive inactivated vaccine, CoronaVac.
  Interventions: Biological: CoronaVac Vaccine

INTERVENTIONS:
Biological: CoronaVac Vaccine — CoronaVac Vaccine
  Groups: CoronaVac
Biological: BNT162b2 Vaccine — Covid-19 BNT162b2 Vaccine
  Groups: BNT162b2

SUMMARY:
Since the first local case of COVID-19 confirmed on 4 Feb 2020, Hong Kong has already experienced 4 waves of COVID-19 surge, with more than 9000 cases reported. A number of vaccines have been shown to be efficacious against symptomatic and severe infection by inducing neutralizing antibody (NAB) against spike protein of the SARS-CoV-2 virus. However, the duration of protection and longevity of antibody response is unknown.

Health care workers (HCWs) who are planning to receive COVID-19 vaccine will be recruited. The level of antibody against spike protein by different quantitative assays will also be serially measured .

ELIGIBILITY:
Inclusion Criteria:

1. Any staff, visiting doctor, nursing student of HKSH who are aged 18 or above
2. No contraindication for COVID-19 vaccination and plan to receive the intended dosages at the appropriate interval.
3. A baseline serology taken within 1 week before vaccination shows no evidence of recent infection.
4. No history of documented COVID-19 infection

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Healthcare workers of HKSH who plan to receive COVID-19 vaccine
Sampling Method: Probability Sample
Enrollment: 480 (Actual)
Dates: Start 2021-03-07 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change of IgG Level in the serum of healthcare workers who received COVID-19 vaccine | 1 month, 3 months and 6 months post vaccination
  Change of IgG Level in the serum of healthcare workers who received COVID-19 vaccine at different points during the first six months of vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Jonpaul Sze Tsing Zee, MBChB, Principal Investigator — Hong Kong Sanatorium & Hotel
Locations (1):
- Hong Kong Sanatorium & Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No